CLINICAL TRIAL: NCT05000632
Title: Establishing Smoke-free Homes With Families Involved in Child Protective Services: Effectiveness-implementation Trial of an Integrated Program
Brief Title: Smoke Free SafeCare: Establishing a Smoke Free Home in CPS-involved Families
Acronym: SFSC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Shannon Self-Brown, Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H21543
Record Dates: First submitted 2021-07-14; First posted 2021-08-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Child Maltreatment; Smoking Behaviors
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at the provider level. Provider participants will be randomized into either Smoke Free SafeCare or Standard SafeCare. Their arm designation will then determine the group that mother participants will be assigned to.
Who Masked: Investigator
Masking Description: Study personnel, including the PI and Co-Is (with the exception of methodologist) and assessment staff, will be masked to treatment condition until the database is locked. Limited staff will be unmasked to handle randomization codes, delivery support of interventions, and to complete reports.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoke Free SafeCare (SFSC) (Experimental): Providers randomized to this group will receive additional SFSC training and will disseminate SFSC program to families who report having a smoker in the home.
  Interventions: Behavioral: Smoke Free SafeCare
- Standard SafeCare (Active Comparator): Providers randomized to this group will disseminate the Standard SafeCare program to families who report having a smoker in the home.
  Interventions: Behavioral: Standard SafeCare

INTERVENTIONS:
Behavioral: Smoke Free SafeCare — SFSC is the systematically braided curriculum which combines both SafeCare and STBO programs, but in a new delivery format. To take full advantage of the home delivery mechanism of SafeCare, the content delivery of STBO has been adapted so that original mailings will be delivered in the SafeCare sessions. STBO has been fully braided into the Health and Safety modules. One of these interventions will be delivered first throughout the course of the study. The Smoke Free SafeCare intervention will involve 25 providers receiving training for the SFSC program. They will each recruit 10 mothers and conduct the SFSC program for each family. Overall, 250 families will receive the SFSC intervention.
  Other Names: SFSC
  Arms: Smoke Free SafeCare (SFSC)
Behavioral: Standard SafeCare — SafeCare is a brief parenting intervention that is highly effective in reducing child maltreatment perpetration and improving behavioral outcomes for CPS-involved parents of young children (0 to 5 years) as the result of child physical abuse or neglect (the two most common forms of substantiated maltreatment). The Standard SafeCare intervention will involve 25 SafeCare providers delivering the SafeCare program as usual. They will each recruit 10 mothers and conduct SafeCare for each family. Overall, 250 families will receive the standard SafeCare.
  Other Names: SafeCare
  Arms: Standard SafeCare

SUMMARY:
Smoke Free SafeCare (SFSC) is a proposed braided intervention consisting of two evidence-based interventions: Some Things are Better Outside (STBO), aimed at promoting smoke free home rules, and SafeCare, aimed at reducing child maltreatment and improving mother and child outcomes. STBO is effective in creating smoke free homes and reducing second-hand smoke in low-SES (socioeconomic status) households. SafeCare is an effective parent training program that is broadly disseminated in child protective services in the United States. SafeCare is a promising mechanism to effectively increase the reach of STBO to reduce SHS (secondhand smoke) exposure in families with documented high rates of tobacco use and children with cumulative risk for negative health outcomes.

DETAILED DESCRIPTION:
Longitudinal studies have found beneficial effects of prevention and intervention efforts for children exposed to poverty and other adverse experiences on long-term health and a range of social and psychological outcomes. Evidence-based intervention programs exist for smoke-free homes and for child maltreatment risk. However, to our knowledge, no programs jointly target SHS (secondhand smoke) exposure and maltreatment risk, despite the evidence that these risk factors often co-occur for children living in low-SES households.

Some Things are Better Outside (STBO) is a brief intervention that is highly effective in promoting adoption of smoke-free home rules among low-SES households. Three randomized controlled trials (RCTs) documented significant intervention effects, with 40.0 to 62.9% of clients reporting a smoke-free home when reached for follow-up at 6 months post-baseline. Self-reported smoke-free homes were validated by air nicotine at 3-months post-baseline. STBO was also effective in a dissemination trial conducted with five 2-1-1 agencies across multiple states. The six-week intervention was designed to be easy to deliver, consisting of three mailings of print materials and a 15-20 minute coaching call.

SafeCare is a brief parenting intervention that is highly effective in reducing child maltreatment perpetration and improving behavioral outcomes for Child Protective Services-involved (CPS-involved) parents of young children (0 to 5 years) as the result of child physical abuse or neglect (the two most common forms of substantiated maltreatment). SafeCare is delivered in the home over 18-weeks, and the curriculum focuses on promotion of positive parenting skills, home safety, and child health. SafeCare is disseminated through the National SafeCare Training and Research Center (NSTRC) at Georgia State University (GSU), directed by Self-Brown (MPI) and Whitaker (Co-I).

In considering the best approaches for targeting SHS, it is imperative to consider how to integrate interventions with documented success for improving smoke-free rules and with high levels of parent engagement (which STBO has consistently demonstrated), into effective parenting intervention programs, such as SafeCare (which has also been demonstrated to be highly engaging). Thoughtful integration would ensure the maintenance of active ingredients for both programs, and parent engagement.

The goal of Smoke Free SafeCare is to conduct an effectiveness-implementation hybrid trial type 1 of the SFSC intervention for parents with substantiated maltreatment. This braided intervention will be compared to standard SafeCare.

The study aims are as follows:

1. To conduct an effectiveness-implementation hybrid trial type 1.
2. Compare SFSC to standard SafeCare on the addition of a full smoking ban in the home, and maintenance and stability of the smoking ban.
3. Understand impact and sustainability of SFSC on parenting outcomes.
4. Examine the variability in SFSC effects across sites and client characteristics.

This project will implement a mixed methods approach to gain insight about the perceived feasibility and impact of SFSC with mothers who report at least two risk factors at initial screening that are commensurate with child maltreatment perpetration risk. Understanding whether there is additive benefit to the integration of these programs will inform policy for best practices of programs serving low-SES families, and will further establish a structured approach for systematically integrating evidence-based programs for populations who have cumulative risk.

ELIGIBILITY:
Provider Inclusion Criteria:

* SafeCare providers in this study must 1) have completed the SafeCare workshop and passed field Certification (9 sessions of SafeCare delivered with fidelity according to the SafeCare Fidelity Checklist); 2) be employed at an accredited SafeCare agency in a target state based on Centers for Disease Control and Prevention (CDC) adult smoking data or prior SafeCare research documenting high smoking rates.

Caregiver Inclusion Criteria:

* Caregivers in this study must meet the following inclusion criteria to participate: 1) Referred to a SafeCare Provider study participant; 2) Reports in-home smoking behavior by herself or another person (person must reside in the home 3 or more nights a week) 3) Caregiver must be aged 18 or older and 4) Mother must be a parent to a child between the ages of 0 and 5 (or 0 - 9 if in the state of Oklahoma).

Provider Exclusion Criteria:

* SafeCare providers will be excluded if they have planned for significant employment leave, resignation, or promotion during the study period.

Caregiver Exclusion Criteria:

* We will exclude those who 1) Report that no one smokes in the home; 2) Demonstrate an inability to understand their responsibilities as outlined in the consent form. This will be determined as the research staff verbally go through the consent form with the mothers. If mothers do not understand the consent form and subsequent procedures, they will be excluded.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Smoke Free Home Rules (Questionnaire) | This outcome will be assessed at baseline.
  Mothers will answer questions specific to smoke free home rules implemented in their home.
Change in Smoke Free Home Rules (Questionnaire) | This outcome will be assessed at the 8 week time point.
  Mothers will answer questions specific to smoke free home rules implemented in their home.
Change in Smoke Free Home Rules (Questionnaire) | This outcome will be assessed at the 20 week time point.
  Mothers will answer questions specific to smoke free home rules implemented in their home.
Change in Smoke Free Home Rules (Questionnaire) | This outcome will be assessed at the 1 year time point.
  Mothers will answer questions specific to smoke free home rules implemented in their home.
Time-Weighted Average Airborne Nicotine - Smoke Free Home Validation | This outcome will be assessed at the 8-week time point.
  Research staff will place an air nicotine monitor in one room in which the family spends the most time. The monitors, the size of a petri dish, will be labeled and left in place for 7 days. For quality assurance and control, one blank sample per 10 samples will be included, along with duplicate samples collected for 10% of the total sample. Research staff will return to the home after 7 days to collect the monitor. Time-weighted average airborne nicotine will be assayed. The amount of nicotine collected is determined in the laboratory using gas chromatographic analysis. The sensitivity of these devices is sufficient to quantify low levels of passive smoke exposures over a period of a few days. Outcome is reported in micrograms of nicotine per cubed meter.
Change in Time-Weighted Average Airborne Nicotine - Smoke Free Home Validation | This outcome will be assessed at the 1 year time point.
  Research staff will place an air nicotine monitor in one room in which the family spends the most time. The monitors, the size of a petri dish, will be labeled and left in place for 7 days. For quality assurance and control, one blank sample per 10 samples will be included, along with duplicate samples collected for 10% of the total sample. Research staff will return to the home after 7 days to collect the monitor. Time-weighted average airborne nicotine will be assayed. The amount of nicotine collected is determined in the laboratory using gas chromatographic analysis. The sensitivity of these devices is sufficient to quantify low levels of passive smoke exposures over a period of a few days. Outcome is reported in micrograms of nicotine per cubed meter.

SECONDARY OUTCOMES:
Parenting Young Children Survey (PYCS) | Assessed at baseline
  Parenting behavior
Parenting Young Children Survey (PYCS) | Assessed at 8-week
  Parenting behavior
Parenting Young Children Survey (PYCS) | Assessed at 20-week
  Parenting behavior
Parenting Young Children Survey (PYCS) | Assessed at 1 year
  Parenting behavior
Perceived Stress Scale | Assessed at baseline
  Measure of personal stress; Min: 0, Max: 5; Higher scores indicated higher perceived stress
Perceived Stress Scale | Assessed at 8 week
  Measure of personal stress; Min: 0, Max: 5; Higher scores indicated higher perceived stress
Perceived Stress Scale | Assessed at 20 week
  Measure of personal stress; Min: 0, Max: 5; Higher scores indicated higher perceived stress
Perceived Stress Scale | Assessed at 1 year
  Measure of personal stress; Min: 0, Max: 5; Higher scores indicated higher perceived stress
Parenting Stress Inventory (PSI) | Assessed at baseline
  Parent stress
Parenting Stress Inventory (PSI) | Assessed at 8-week
  Parent stress
Parenting Stress Inventory (PSI) | Assessed at 20 week
  Parent stress
Parenting Stress Inventory (PSI) | Assessed at 1 year
  Parent stress
Smoking Cessation Questionnaire | Assessed at baseline
  These questions assess parents attempts to stop or minimize smoking behaviors
Smoking Cessation Questionnaire | Assessed at 8-week
  These questions assess parents attempts to stop or minimize smoking behaviors
Smoking Cessation Questionnaire | Assessed at 20-week
  These questions assess parents attempts to stop or minimize smoking behaviors
Smoking Cessation Questionnaire | Assessed at 1 year
  These questions assess parents attempts to stop or minimize smoking behaviors

OTHER OUTCOMES:
Demographic - Number of Children | This item may change over time so it will be assessed at baseline, 8-week, 20-week, and 1-year (i.e. employment status, number of children, etc.)
  Number of Children at the time of assessment
Demographic - Employment Status | This item may change over time so it will be assessed at baseline, 8-week, 20-week, and 1-year (i.e. employment status, number of children, etc.)
  Employment status at the time of assessment
Demographic - Age | This item may change over time so it will be assessed at baseline, 8-week, 20-week, and 1-year (i.e. employment status, number of children, etc.)
  Age at time of assessment
Demographic - Sex assigned at birth | Assessed at baseline
  Sex assigned at birth
Demographic - Gender | Assessed at baseline
  Gender
Demographic - Race | Assessed at baseline
  Race
Demographic - Ethnicity | Assessed at baseline
  Ethnicity
Demographic - Relationship status | This item may change over time so it will be assessed at baseline, 8-week, 20-week, and 1-year (i.e. employment status, number of children, etc.)
  Relationship status at time of assessment
Demographic - Education | Assessed at baseline
  Highest grade/level completed in school
Demographic - Disability | This item may change over time so it will be assessed at baseline, 8-week, 20-week, and 1-year (i.e. employment status, number of children, etc.)
  Supported by disability at time of assessment
Demographic - Household income | This item may change over time so it will be assessed at baseline, 8-week, 20-week, and 1-year (i.e. employment status, number of children, etc.)
  Household income at time of assessment

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Self-Brown, PhD, Principal Investigator — Georgia State University; Michelle Kegler, Principal Investigator — Emory University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data related to a dataset on parent and implementation outcomes have the potential to be shared with other researchers, if requested.
Supporting Information: SAP, CSR, Analytic Code
Time Frame: IPD sharing will occur once the study is complete and will continue for up to two years after study completion.
Access Criteria: Resource Sharing: This research will generate a dataset on parent and implementation outcomes for Smoke-Free SafeCare in child welfare settings in at least two states. If an investigator who is not part of our collaborative team requests these data, we will in turn request a research proposal that describes his/her research question, which variables/codes she/he would like to use, analysis plans, and proposed dissemination plans. Our investigator team will review and make decisions about these requests. Once we have completed our primary analyses, we will upload the de-identified quantitative datasets to an online data storage site, with accompanying documentation.

REFERENCES:
- [Derived] Perry EW, Self-Brown S, Koontz K, Haardorfer R, Whitaker DJ, Spears CA, Huang J, Kegler M. Evaluating the effectiveness of Smoke-Free Home SafeCare, an integrated intervention, among families at risk for secondhand smoke exposure and child maltreatment in the United States: a study protocol for a hybrid type 1 trial. Trials. 2024 Oct 7;25(1):661. doi: 10.1186/s13063-024-08466-2. PMID 39375710
- [Derived] Self-Brown S, Perry EW, Recinos M, Cotner MA, Guastaferro K, Owolabi S, Spears CA, Whitaker DJ, Huang J, Kegler MC. Systematic braiding of Smoke-Free Home SafeCare to address child maltreatment risk and secondhand smoke exposure: findings from a pilot study. Pilot Feasibility Stud. 2023 May 12;9(1):81. doi: 10.1186/s40814-023-01303-4. PMID 37173799